CLINICAL TRIAL: NCT04678141
Title: Clinical Evaluation of Compomer and Composite Class II Restorations in Primary Molars: 24 Months Results
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Suleyman Demirel University (Other)
Responsible Party: Principal Investigator, Esra Oz, Assistant professor, Suleyman Demirel University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 72867572.050.01.04-207321
Record Dates: First submitted 2020-12-10; First posted 2020-12-21 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Primary Teeth
Keywords: class II; compomer; composite resin; primary molars; restoration

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Composite and compomer materials (Other): Children aged 5-6 years with at least two carious proximal surface primary molars
  Interventions: Other: Dyract XP (Dentsply De Trey), Kerr Herculite Classic (Kerr Corporation),R&D Series NOVA(Kuraray Medical Inc) Clearfil TM SE Bond (Kuraray Medical),Hydrocal LC (Medicept Dental)

INTERVENTIONS:
Other: Dyract XP (Dentsply De Trey), Kerr Herculite Classic (Kerr Corporation),R&D Series NOVA(Kuraray Medical Inc) Clearfil TM SE Bond (Kuraray Medical),Hydrocal LC (Medicept Dental) — compomer (Dyract XP,R&D Series NOVA) , composite (Kerr Herculite Classic),Bonding (Clearfil TM SE Bond), Dycall (Hydrocal LC)

SUMMARY:
It was aimed to evaluate the clinical performance of resin-hybrid composite and compomer materials in primary molars over a 2-year period.

DETAILED DESCRIPTION:
All treatment stages were performed by the same experienced pediatric dentist (E.O.) to avoid behavioral problems. When necessary, topical anesthesia with 2% Xylocaine® DENTAL was administered, followed by local anesthesia with epinephrine 1: 100.000 (lidocaine HCl and Epinephrine Injection, DENTSPLY Pharmaceutical, USA). Access to proximal surfaces was provided with high-speed diamond bur (FD.D.801, Frank Dental, Germany) under an air-water coolant. The proximal cavity was opened at the occlusal level. Soft carious dentine was removed with a round low-speed steel bur (SS.1A, Frank Dental, Germany).

Restorations were placed under isolation with cotton rolls and a saliva ejector. The Ca(OH)2 cavity liner material (Hydrocal LC, Medicept Dental, India) was used as base material if the distance from the pulp was not safe. A metal matrix band (Matrix band, Hahnenkratt, Königsbach-Stein, Germany) was applied to the tooth with a universal matrix system (Tofflemire, Hahnenkratt, Königsbach-Stein, Germany) and wooden wedges (TDV, No 1). ClearfilTM SE Bond (Kuraray Medical Inc, Okayama, Japan) was applied to the cavity according to the manufacturer's instructions. For the polymerization, an LED curing light (Eliapar Freelight, 3M ESPE Dental Products, America) was used with a light power density of 600 mW/cm2. According to the manufacturer's instructions, A2 composite resin (Kerr Herculite Classic) and two different compomer materials (Dyract/XP and R&D Series NOVA) were applied to the teeth with the incremental technique, and each increment was light-polymerized for 20 sec with an LED curing light.

ELIGIBILITY:
Inclusion Criteria:

* Mentally and physically healthy

Exclusion Criteria:

* Systemic disease or medical complications

Ages: 5 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 145 (Actual)
Dates: Start 2018-07-23 (Actual); Primary Completion 2018-10-23 (Actual); Study Completion 2020-08-23 (Actual)

PRIMARY OUTCOMES:
USPHS criteria | up to 2 years
  Clinical evaluation of composite resin and compomer restorations in primary molars

CONTACTS AND LOCATIONS:
Overall Officials: Esra Oz, Assist Prof, Study Director — Suleyman Demirel University
Locations (1):
- Suleyman Demirel University Faculty of Dentistry Pediatric Dentistry Department, Isparta, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Tseveenjav B, Furuholm J, Mulic A, Valen H, Maisala T, Turunen S, Varsio S, Auero M, Tjaderhane L. Survival of extensive restorations in primary molars: 15-year practice-based study. Int J Paediatr Dent. 2018 Mar;28(2):249-256. doi: 10.1111/ipd.12348. Epub 2017 Dec 3. PMID 29205613
- [Result] Chisini LA, Collares K, Cademartori MG, de Oliveira LJC, Conde MCM, Demarco FF, Correa MB. Restorations in primary teeth: a systematic review on survival and reasons for failures. Int J Paediatr Dent. 2018 Mar;28(2):123-139. doi: 10.1111/ipd.12346. Epub 2018 Jan 10. PMID 29322626
- [Result] Fuks AB. The use of amalgam in pediatric dentistry: new insights and reappraising the tradition. Pediatr Dent. 2015 Mar-Apr;37(2):125-32. PMID 25905653
- [Result] Fuks AB, Araujo FB, Osorio LB, Hadani PE, Pinto AS. Clinical and radiographic assessment of Class II esthetic restorations in primary molars. Pediatr Dent. 2000 Nov-Dec;22(6):479-85. PMID 11132507